CLINICAL TRIAL: NCT04689139
Title: Role of Intraoperative Biomarkers in Prognosis of Perioperative Complications in Reconstructive Thoracic Aorta Surgery
Brief Title: Biomarkers in Thoracic Aorta Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 039420200002
Record Dates: First submitted 2020-12-22; First posted 2020-12-30 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Aortic Aneurysm; Thoracoabdominal Aneurysm; Aortic Dissection; Complication
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thoracic aorta surgery patients (Experimental): Blood samples on proadrenomedullin, presepsin, NT-proBNP, Troponin I, procalcitonin are acquired
  Interventions: Diagnostic Test: blood sample tests for determination of biomarkers levels

INTERVENTIONS:
Diagnostic Test: blood sample tests for determination of biomarkers levels — Using of proadrenomedullin, presepsin, NT-proBNP, Troponin I to determine the correlation of perioperative complications.

SUMMARY:
Biomarkers can play a vital role in prognosing the perioperative complications in thoracic aorta surgery. The goal of a study is to determine the correlation between intraoperative level of certain biomarkers and total amount of peroperative complications.

DETAILED DESCRIPTION:
This study aims to assess the association between levels of biomarkers and postoperative complications in patients after thoracic and thoracoabdominal aortic reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Elective thoracic and thoracoabdominal surgery

Exclusion Criteria:

* Hemolysis in blood sample

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Akselrod, Professor, Study Director — Petrovsky NRCS
Locations (1):
- Petrovsky Research National Centre of Surgery ( Petrovsky NRCS), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Assessing the significance of some biomarkers in perioperative period after thoracic aortic reconstruction — https://russjcardiol.elpub.ru/jour/article/view/5314/4231

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thoracic Aorta Surgery Patients
Started | 132
Completed | 132
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Thoracic Aorta Surgery Patients
Number analyzed (Participants) | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 132
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 132
Body surface area, м² [Mean (Standard Deviation); unit: square meters] | 2 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: Number of Total Postoperative Complications
Description: Value reported in the Outcome Measure data table reflects the Number of Total Postoperative Complications across all participants.
Time Frame: up to 10 days
Measure: Number; unit: post-operative complications
Arm/Group | Thoracic Aorta Surgery Patients
Number analyzed (Participants) | 132
post-operative complications | 69

2. Secondary Outcome: Total Number Affected by All-Cause Mortality
Description: Overall number of participants, in each arm/group, who died due to any cause
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Aorta Surgery Patients
Number analyzed (Participants) | 132
Participants | 2

3. Secondary Outcome: Number of Participants Who Require Extracorporeal Detoxication
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Aorta Surgery Patients
Number analyzed (Participants) | 132
Participants | 7

4. Secondary Outcome: Number of Cardiac Disorders
Description: Number of patients who needed medicamental cardiotonic support more than 1 day
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Aorta Surgery Patients
Number analyzed (Participants) | 132
Participants | 16

5. Secondary Outcome: Number of Vascular Disorders
Description: Number of patients who needed vasopressor support more than 1 day
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Aorta Surgery Patients
Number analyzed (Participants) | 132
Participants | 14

6. Secondary Outcome: Number of Infections and Infestations
Description: Number of patients who develop systemic infection and/or operation wound infection
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Aorta Surgery Patients
Number analyzed (Participants) | 132
Participants | 36

ADVERSE EVENTS:
Time Frame: Up to 10 days postoperative
Arm/Group | Thoracic Aorta Surgery Patients
All-Cause Mortality (participants affected / at risk) | 2/132
Serious Adverse Events (participants affected / at risk) | 41/132
Other Adverse Events (participants affected / at risk) | 24/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thoracic Aorta Surgery Patients (N=132)
Patients requiring extracorporeal detoxication (Renal and urinary disorders) | 7 (7)
Pneumonia (Infections and infestations) | 29 (29)
Myocardial infarction (Cardiac disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thoracic Aorta Surgery Patients (N=132)
Cardiac dysrhythmias (Cardiac disorders) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT04689139/Prot_SAP_001.pdf